CLINICAL TRIAL: NCT04991688
Title: A Prospective Pilot Study to Assess the Efficacy of Botox-A in Patients With Low Anterior Resection Syndrome (LARS>20) and Refractory Medical Treatment After Rectal Resection
Acronym: BOTOX-TME
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Organizational difficulties
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2020/64
Record Dates: First submitted 2021-06-25; First posted 2021-08-05 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Low Anterior Resection Syndrome (LARS>20); Refractory Medical Treatment After Rectal Resection
Keywords: Rectal surgery; Low Anterior Resection syndrome; Refractory medical treatment; Fecal incontinence
MeSH Terms: conditions — Low Anterior Resection Syndrome; Fecal Incontinence | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BOTOX-A (Experimental)
  Interventions: Drug: BOTOX-A

INTERVENTIONS:
Drug: BOTOX-A — 10 injections of 20 U of toxin will be made into the rectum 5, 10 and 15 cm above the pectinate line. At each level, 3 injections of 20 U will be performed in the submucosa, circumferentially.The last injection is made 20 cm above the pectinate line. Total does not exceed 200U of Botox-A

SUMMARY:
After rectal resection for cancer (with or without stoma), patients may have digestive sequelae. LARS (Low Anterior Resection Syndrome) includes bowel frequency, stool fragmentation, urgency, and faecal incontinence. The goal of this study is to test intra-rectal BOTOX-A on functional outcomes and quality of life of patients with LARS refractory to medical treatment at 3 months after surgery.

DETAILED DESCRIPTION:
Bowel dysfunction after low anterior resection (rectal excision) is referred as Low Anterior Resection Syndrome (LARS). LARS includes bowel frequency, stool fragmentation, urgency, and faecal incontinence. LARS negatively affects patients' quality of life by impacting emotional, physical, social, and role functioning. Symptoms may persist up to 15 years after surgery.

The treatment options for LARS include successively conservative options, as medical drugs and biofeedback, and aggressive options, as retrograde colonic washout, sacral neuromodulation, antegrade colonic enema via a caecostomy, or a definitive colostomy. The effectiveness of conservative treatment remains uncertain and the aggressive treatments are associated with daily constraints and potential morbidity. These findings highlight the need for more efficient treatments BOTOX-A is a neurotoxin inhibiting acetylcholine release at the neuromuscular junction. BOTOX-A has displayed significant benefits in patients with urinary incontinence, demonstrating significant efficacy as compared to placebo. Intra-rectal injections of Botox-A has been trialed for the treatment of over active rectum induced fecal incontinence. Improvement of symptoms and quality of life have been demonstrated. Currently an ongoing national multicenter trial in France, IF Toxine (N° CLINICAL TRIAL: NCT02414425), has included 200 patients to assess Botox-A intra-rectal injections as a treatment option for fecal incontinence, without any safety concerns observed.

The investigators anticipate that BOTOX-A injections could represent a medical option to treat digestive dysfunction (LARS) after surgery for rectal cancer, by reducing the spasm of the smooth muscle in the colon working as a neorectum.

Globally 50% of patients were refractory to medical treatment (LARS score > 20) at 3 months after surgery. Of those, only 30% of them were improved by prolonged medical treatment between 3 and 6 months. The investigators anticipate that 60 % of them will be improved by association of medical treatment and BOTOX-A injection.

The objective is to assess the efficacy of BOTOX-A on the proportion of patients with bowel dysfunction (LARS score > 20) at 3 months after injection.

ELIGIBILITY:
Inclusion Criteria:

* Patient: male and female, age ≥18 years
* Tumour: rectal cancer
* Surgery: anterior resection (high or low) with colorectal or coloanal anastomosis, or intersphincteric resection, or pull-through
* Symptoms: Low Anterior Resection Syndrome (LARS score >20) refractory to medical treatment at 3 months after rectal surgery (or after temporary stoma closed)
* Straight or pouch colonic reconstruction
* Surgery alone or with neoadjuvant therapy (chemoradiotherapy, short course radiotherapy, induction chemotherapy)
* Signed and dated informed consent
* Patient affiliated to a social security system or beneficiary of the same
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures

Exclusion Criteria:

* Anal cancer
* Anal surgery in the last 3 months
* Acute/painful perianal disease
* Ongoing adjuvant treatment
* Contraindication for BOTOX-A (known hypersensitivity to botulinum toxin type A or to albumin, infection at the proposed injection site, severe myasthenia)
* Have received BOTOX-A in perianal region in the previous 3 months
* General anesthesia performed less than a month
* Impossibility of performing a rectoscopy (eg: anal stenosis)
* Recent history (<12 months) of myocardial infarction and / or arrhythmias not reduced by appropriate treatment
* Subject with a significant deficit of clinical or subclinical neuromuscular transmission (myasthenia or Lambert-Eaton syndrome) or with peripheral motor neuropathy (such as amyotrophic lateral sclerosis or motor neuropathy)
* Treatment that directly or indirectly interferes with neuromuscular transmission (aminoglycosides, curare, anticholinesterase, aminoquinoline, cyclosporine, etc.)
* History of neuromuscular disorders
* Anal clinical examination suggesting the presence of an anorectal abscess
* Pregnant woman or breastfeeding woman
* Women of child-bearing potential (WOCBP)* not using effective contraception (oestrogen-progesteron combined contraceptives or intra uterine device) since at least 7 days and during all the duration of the study
* Persons deprived of their liberty or under measure of judicial protection (curatorship or guardianship) or unable to give their consent
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol or follow-up schedule, as assessed by investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-01-07 (Actual); Study Completion 2023-03-03 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with LARS > 20 | At 3 months after injection

SECONDARY OUTCOMES:
Compliance to treatment | At 3 months after injection
  Proportion of patients receiving full injections, 10 injections of 20U of toxin. A total of 200U of BOTOX A will be injected
Tolerance to treatment | At 3 months after injection
  Number of patients with adverse events
Functional outcome with LARS score | At 0, 1, 2, 3 and 6 months
  The LARS questionnaire (Low Anterior Resection Syndrome) was the primary end-pointy and evaluate bowel function. Five questions regarding incontinence for flatus and liquid stools, frequency, clustering and urgency for defecation are taken into account. The score ranges from 0 to 42 is divides into no LARS (0 to 20 points), minor LARS (21 to 29 points), and major LARS (30 to 42 points)
Faecal incontinence with Wexner score | At 0, 1, 2, 3 and 6 months
  The Wexner score assesses the importance of anal incontinence, it varies from 0 to 20, 20 corresponding to total incontinence
Quality of life (QLQ C-30) | At 0, 1, 3 and 6 months
  The scores of questionnaire QLQ C-30 will be examined
  The EORTC QLQ-C30 is a patients self-rating questionnaire that measures physical, role, social, emotional, and cognitive functions as well as overall QoL. Scores can be linearly transformed to provide a score from 0 to 100. Higher scores represent better functioning on the functional scales and a higher level of symptoms of the symptom scales.
Quality of life (QLQ CR-29) | At 0, 1, 3 and 6 months
  The scores of questionnaire QLQ CR-29 will be examined
  The EORTC QLQ-CR29 has five functional and 18 symptom scales. Scores can be linearly transformed to provide a score from 0 to 100. Higher scores represent better functioning on the functional scales and a higher level of symptoms of the symptom scales.
Evaluation of Anxiety profil (STAI-Y : State-Trait Anxiety Inventory ) | At 0, 1, 3 and 6 months
  For evaluation of Anxiety profil , the "state" instructions is used, which require participants to report how they feel "right now, at this moment," and the "trait" instruction, which ask them to indicate how they "generally"feel. . For each subscales, scores range from 10 to 40, with higher scores correlating with greater state or trait anxiety.
Evaluation of manometry | At 0, 1, 3 and 6 months
  Manometry will measure the pressure in mmHg of the ano-rectal passage, specifically pressures corresponding to the internal and external sphincter, and rectum. The resting pressure and squeeze pressure will be assessed. Sensitivity test to assess first sensation of gas, urge to defecate, and urgency will also be assessed.
Evaluation of barostat | At 0, 1, 3 and 6 months
  Barostat allows the measurement of rectal capacity (ml) and compliance (ml/mmHg). Compliance is a dynamic property of the rectum, calculated from a sigmoid curve of pressure vs volume created by a step wise incremental distention sequence of a balloon placed in the rectum. Compliance of the patient population (post TME surgery) can be compared to compliance of non-operated rectums from published data. The investigators anticipate that our patient population will have a less compliant neo-rectum and hope to see a difference after Botox-A injection
Proportion of patients with LARS ≤ 20 | At 6 months
Correlation between LARS and physiologic tests | At 0, 1, 2, 3 and 6 months
  The correlation of objective physiologic measures such as manometry and barostat will be compared and correlated to the symptoms described by the patient in the LARS questionnaire before and after injection of Botox-A in the neo-rectum.The investigators anticipate a correlation of increased compliance in the neo rectum with improvement of symptoms (lower LARS score) post Botox-A injection

CONTACTS AND LOCATIONS:
Overall Officials: Eric RULLIER, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- CHU Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No